CLINICAL TRIAL: NCT05401708
Title: A Prospective Cohort Study for Establishing Clinical Excellence in Patients With Newly Diagnosed Type 1 and Type 2 Diabetes and Prediabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0234
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Newly Diagnosed Type 1 and Type 2 Diabetes and Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Preservation of urinary samples: After performing conventional urinary tests, the residual urinary samples are collected. Samples are centrifuged and supernatant of each sample (5mL) is subdivided into 1mL into cryotube (total 5 cryotubes for preservation), which are deep frozen in -80℃. (In order to avoid problems caused by freezing-thawing process, researchers decided to subdivide sample) These 5 samples will be registered for further evaluations.
  * Preservation of blood samples: After performing conventional blood tests, the residual or additional blood samples are collected. Samples are centrifuged and serum of each sample is subdivided into 1mL into cryotube (total 10 cyrotubes for preservation), which are deep frozen in
  * 70℃ or liquid nitrogen tank. These 10 samples will be registered for further evaluations.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DM Naïve: a new patient without a history of DM medication

SUMMARY:
Diabetes mellitus is recognized as a metabolic disease that causes global economic and health burdens with an estimated number of patients 135 million in 1995 to 300 million in 2025. Moreover, the Asia-Pacific region is considered to be on the verge of an emerging diabetes epidemic. Diabetes is associated with numerous comorbidities due to a wide range of complications, such as retinopathy, nephropathy, neuropathy, and cardiovascular disease, which could lead to premature mortality. Management of diabetes under standard treatment protocol improves quality of life and prevents complications and premature mortality. Pathogenesis of these detrimental complications caused by diabetes is not yet discovered and it is important to reveal epidemiology and mechanisms of diabetes and its complications in order to successfully manage and control diabetes. According to the Committee of the Korean Diabetes Association on the Epidemiology of Diabetes Mellitus, only about one third of patients with diabetes was found to reach target glycemic control (<7% of HbA1c) and 30.3%, 38.3% and 44.6% of patients found to have microalbuminuria, retinopathy and nephropathy, respectively in tertiary hospitals of Korea in 2006. Also, prevalence of coronary artery disease, cerebrovascular disease and peripheral artery disease was 8.7%, 6.75 and 3.0%, respectively in tertiary hospitals. Due to inadequate achievement of glycemic control and improper prevention tactics to prevent diabetic complication for patients in tertiary hospitals in Korea, it is pivotal to determine and analyze the current status of patients with diabetes and prediabetes for efficient management of diabetes/prediabetes and its complications. Annual visits of newly diagnosed diabetes or prediabetes to Endocrinology department of Severance hospital in Korea are increasing, about 5,000 patients per year since 2017. However, there is no current systemic clinical registry involving patients with diabetes or prediabetes in Severance hospital. Therefore, in this prospective cohort study, we will establish registry for patients with diabetes or prediabetes who would perform standard blood/urine tests and follow treatment protocols in Endocrinology department of Severance hospital.

ELIGIBILITY:
Inclusion Criteria:

* Drug naive patients who are newly diagnosed type 1 diabetes/type 2 diabetes or prediabetes since March, 2022 in Severance hospital ② Male or female who are older than 20 years ③ Patients who consented and underwent recommended regular blood and urinary tests according to the current guidelines.

Exclusion Criteria:

① Patients who are considered to be unable to participate in the study by the judgement of researchers

② Patients who are unable to read the consent forms (E.g Foreigner, illiteracy)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited Severance hospital from March, 2022 with newly diagnosed type 1 diabetes/type 2 diabetes or prediabetes and consented and underwent regular blood and urinary tests acccording to the current guidelines Inclusion criteria
  * Drug naive patients who are newly diagnosed type 1 diabetes/type 2 diabetes or prediabetes since March, 2022 in Severance hospital ② Male or female who are older than 20 years ③ Patients who consented and underwent recommended regular blood and urinary tests according to the current guidelines.
  Exclusion criteria ① Patients who are considered to be unable to participate in the study by the judgement of researchers
  ② Patients who are unable to read the consent forms (E.g Foreigner, illiteracy)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood and urinary tests and complications in patients with type 1 and 2 diabetes mellitus and prediabetes (cross-sectional) | Annually for 5 years.
  Blood and urinary samples : fasting glucose/insulin/c-peptide, HbA1c, glycoalbumin, beta-hydroxybutyrate, free fatty acid-fasting, postprandial 90 min glucose/insulin/c-peptide, BUN, creatinine, eGFR, AST, ALT, ALP, GGT, total bilirubin, total protein, albumin, uric acid, total cholesterol, triglyceride, HDL, LDL, WBC, RBC, hemoglobin, hematocrit, platelet, c-reactive protein, urine Glucose, Creatinine, Microprotein, total, Microalbumin, Urinalysis with Microscopy, Urinary N-acetyl beta-D glucosaminidase Complication study: Liver Fibroscan, fundoscopy, Intima media thickness, Nerve conduction velocity, Fat u/s & Body Index, Pulse wave velocity & ankle brachial index, Autonomic nervous system

CONTACTS AND LOCATIONS:
Overall Officials: BYEONGWAN LEE, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No